CLINICAL TRIAL: NCT05201768
Title: Determination of Walking, Balance, Fall Risk and Kinesiophobia in Individulas with Alzheimer's Dementation
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Oguzhan Dogancı, Physiotherapist, Kırıkkale University
Other Study IDs: kku-oguzhandoganci1
Record Dates: First submitted 2021-12-07; First posted 2022-01-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- INDIVIDUALS WITH ALZHEIMER: balance and gait will be evaluated survey questions will be asked
  Interventions: Other: balance tests,questionnaire
- HEALTHY INDIVIDUALS: balance and gait will be evaluated survey questions will be asked
  Interventions: Other: balance tests,questionnaire

INTERVENTIONS:
Other: balance tests,questionnaire — Individuals will be tested and recorded.

SUMMARY:
THE OBJECTIVE OF THE RESEARCHERS IS TO DETERMINE WALKING, BALANCE, FALL RISK AND KINESIOPHOBIA IN INDIVIDUALS WITH ALZHEIMER'S DEMENTATION.

DETAILED DESCRIPTION:
The gait, balance, fall risks and kinesiophobia of individuals with Alzheimer's Dementia will be evaluated and compared with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* INDEPENDENT walker diagnosed with Alzheimer's Dementia

Exclusion Criteria:

* Having a disability to do physical activity Those who have had an operation in the last 6 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 36 individual
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Age | 5 month
  between the ages of 50 and 80
Body Mass Index | 5 month
  BMI was recorded in kg/m^2

SECONDARY OUTCOMES:
The Tinetti Gait and Balance Test (TGBT) | 5 month
  TGBT consists of balance and gait subheadings. For balance, there are 13 items, and 9 items for gait. Items are scored as 0 (abnormal), 1 (adaptive) and 2 (normal) for balance, 0 (abnormal), 1 (normal) for gait. The maximum balance score of the patient is 26 and the maximum gait score is 9. Total score (balance + walking) is 35 points.
Mini Mental State Test | 5 month
  It was used to determine the cognitive state before the training. The Mini-Mental State Test was first published by Folstein et al. It consists of eleven items under 5 main headings: orientation, record memory, attention and calculation, recall and language, and the total score is evaluated over 30 points.
Tampa Scale | 5 month
  17 questions is a scale. The scale is used in work-related activities, injury/re-injury and fear-avoidance contains the parameters.
The Time Up Go Test | 5 month
  The timed "Up & Go" measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm), walk a distance of 3 meters, turn, walk back to the chair, and sit down again.
The Gait Speed Measurement Test (GSMT) | 5 month
  For GSMT, individuals were asked to walk at a speed they wanted on a flat surface of 14 m. Signs were placed on the 2nd and 12th meters of the test area to minimize the speed changes between walking start and walking finish, and to make a more objective measurement. The walking time at this 10-meter distance was measured with the stopwatch and the results were recorded in sec and the walking speed was determined.
Fall Risk Self-Assessment Scale | 5 month
  It consists of 13 items assessing the risk of falling in the elderly. The answers are yes (1 point) and no (0 points), and individuals who get 4 points or more from the scoring are classified as having a high risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuzhan Doğancı, Study Chair — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
test results of individuals, information such as height and weight will be published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1.03.2022-1.07.2022
Access Criteria: open access

REFERENCES:
- [Derived] Doganci O, Sertel M. Determination of balance, fall risk, and kinesiophobia in individuals with Alzheimer's Dementia. Front Psychol. 2025 Mar 11;16:1535440. doi: 10.3389/fpsyg.2025.1535440. eCollection 2025. PMID 40134734